CLINICAL TRIAL: NCT03135353
Title: Comparison Between 3D Saline Infusion Sonohystrography and Office Hysteroscopy in the Evaluation of Patients With Irregular Uterine Bleeding
Brief Title: Saline Sonohystrography and Office Hysteroscopy in Evaluation of Cases of Abnormal Uterine Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, Assistant Professor Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: ED200417
Record Dates: First submitted 2017-04-20; First posted 2017-05-01 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D saline infusion sonohysterography (Experimental): participants presenting with abnormal uterine bleeding will undergo 3D saline infusion sonohysterography
  Interventions: Device: 3D saline infusion sonohysterography
- Office hysteroscopy (Experimental): after undergoing 3D SIS, cases would undergo office hysteroscopy and the investigator would be blinded to the results of SIS
  Interventions: Device: Office Hysteroscopy

INTERVENTIONS:
Device: 3D saline infusion sonohysterography — instillation of saline in the uterine cavity using pediatric foley's catheter, then performing 3D ultrasound scan of the uterus and adenexae
  Arms: 3D saline infusion sonohysterography
Device: Office Hysteroscopy — an outpatient procedure done to assess the uterine cavity using the office hysteroscopy
  Arms: Office hysteroscopy

SUMMARY:
comparing the efficacy of the 3D saline infusion sonohysterography to the diagnostic office hysteroscopy in the diagnosis of the cause of abnormal uterine bleeding in females during their reproductive age

ELIGIBILITY:
Inclusion Criteria:

* female aged between 20 and 45 years
* with no medical disorders
* approving to participate in the study

Exclusion Criteria:

* vaginal or cervical lesions
* history or suspicion of PID
* IUD users
* bleeding disorders
* on anticoagulant therapy
* irregular use of oral contraceptive pills

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-11-25 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
effectiveness of SIS versus office hysteroscopy in the diagnosis of cause of AUB | 6 months
  The results of the two procedures would be compared with the operative findings and later histopathological assessment of the specimens

CONTACTS AND LOCATIONS:
Overall Officials: Dina MR Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el ainy hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No